CLINICAL TRIAL: NCT05163886
Title: A Phase IIa Trial to Evaluate the Safety, Tolerability, and Biological Activity of LAM-002A (Apilimod Dimesylate Capsules) in C9ORF72-Associated Amyotrophic Lateral Sclerosis
Brief Title: Study of Safety, Tolerability, and Biological Activity of LAM-002A in C9ORF72-Associated Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAM-002A-ALS-CLN01
Record Dates: First submitted 2021-11-17; First posted 2021-12-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-09

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: C9ORF72
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LAM-002A (Experimental): LAM-002A will be administered orally in five 25 mg capsules twice a day (250 mg total daily dose).
  Interventions: Drug: LAM-002A
- Placebo (Placebo Comparator): Placebo matching LAM-002A will be administered orally in 5 capsules twice a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LAM-002A — LAM-002A (apilimod dimesylate) is formulated in capsules containing 25 mg of apilimod dimesylate. The capsule is Swedish orange, size 0.
  Arms: LAM-002A
Other: Placebo — Microcrystalline cellulose in Swedish orange, size 0 capsules.
  Arms: Placebo

SUMMARY:
This is a clinical trial to evaluate the safety, tolerability, and biological effect of LAM-002A in adults with C9ORF72-associated ALS (C9ALS).

DETAILED DESCRIPTION:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, biomarker-driven clinical trial evaluating the safety, tolerability, and biological effect of LAM-002A in approximately 12 adults with C9ORF72-associated ALS (C9ALS).

In Part A of the study, approximately twelve C9ALS participants will receive either standard of care plus LAM-002A or standard of care and placebo (randomized 2:1) for the first 12 weeks of the study (Core Study). LAM-002A will be administered as oral capsules 125 mg BID (250 mg total daily dose). The LAM-002A dose may be reduced to 100 mg BID (200 mg total daily dose) if expected gastrointestinal side effects develop.

Participants who complete the first 12 weeks of the Core Study will be eligible to receive active drug (LAM-002A capsules at maximum tolerated dose of 125 or 100 mg BID) for the remainder of the study (open-label extension [OLE]) up to Week 24.

In Part B of the study, participants who complete Part A Week 24 on study drug, will be offered the opportunity to opt-in to continue the open label extension for additional 36 weeks starting at the week 24 visit. Participants who elect not to roll over into the Treatment period B will complete the Day 168 visit, followed a final safety telephone call visit at week 28 to complete study participation. Participants who opt-in to the open label extension for an additional 36 weeks will have their end of study safety telephone call at week 64.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of C9ORF72-associated ALS with BOTH of the following:

   1. Documentation of a clinical genetic test demonstrating the presence of a pathogenic repeat expansion in C9ORF72. If there is a strong clinical suspicion for C9ALS based on C9-positive family history and El Escorial Criteria consistent with a diagnosis of ALS, clinical testing for the C9ORF72 repeat expansion may be performed with study screening labs at the discretion of the Site Investigator (SI), medical monitor, and study sponsor.

      AND
   2. Must meet possible, laboratory-supported probable, probable, or definite criteria for diagnosing ALS by revised El Escorial criteria (Brooks 2000).
2. Age 18 or older
3. Capable of providing informed consent at the Screening Visit and complying with study procedures throughout the study, in the SI's opinion, and at the discretion of the medical monitor and study sponsor.
4. In the case that a participant lacks the ability to provide informed consent. Informed consent will be sought from the participant's surrogate representative.
5. Able to safely swallow study drug capsule at screening and throughout study. May use thickened substances to assist in swallowing drug.
6. Vital Capacity greater than and equal to 50% of predicted at the time of the Screening Visit measured by Slow Vital Capacity (SVC), or, if required due to COVID-19 pandemic-related restrictions and with Sponsor approval, Forced Vital Capacity (FVC) measured in-person or via telemedicine.
7. Participants must either not take or be on a stable dose of riluzole (as either a tablet or oral suspension) for greater than 30 days prior to the Screening Visit. Riluzole-naïve participants are permitted in the study.
8. Participants must either not take edaravone or have completed at least one 14-day cycle with plan for continuation of edaravone prior to the Screening Visit. Participants must be off cycle and at least 2 days after the last dose administration of edaravone at the time of study visit. Edaravone-naïve participants are permitted in the study.
9. Participants must be able to complete all study procedures, including the lumbar punctures (LP) at the time of the Screening Visit, in the SI's opinion.
10. Geographically accessible to the site.

Exclusion Criteria:

1. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant, according to the SI's judgment [e.g., cardiovascular instability, systemic infection, or clinically significant laboratory abnormality or electrocardiogram (ECG) changes].

   1. Gastrointestinal disease (e.g., gastric, or intestinal bypass surgery, jejunostomy tube, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction) that might interfere with drug absorption or with interpretation of gastrointestinal AEs. Gastrostomy tube placement is allowed prophylactically or to supplement nutrition/hydration but may not be used for study drug administration.
   2. Hepatic profile showing any of the following:

   i. Serum alanine aminotransferase (ALT) greater than 5 × upper limit of normal (ULN).

   ii. Serum aspartate aminotransferase (AST) greater than 5 × ULN.

   iii. Serum bilirubin greater than 1.5 × ULN.

   c. Renal profile showing an estimated creatinine clearance (eClCR) less than 30 mL/minute (with eClCR to be calculated by the method at the laboratory performing the serum creatinine test).
2. Presence of a neurodegenerative cognitive or motor syndrome (e.g., Alzheimer's disease, Parkinson's disease) not related to the C9ORF72 repeat expansion.
3. Presence of unstable psychiatric disease or substance abuse that would impair ability of the participant to provide informed consent, in the SI's opinion.
4. Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years. Active cancer includes cancers with current disease manifestations or therapy that could adversely affect subject safety and longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
5. Prior solid organ transplantation.
6. Ongoing immunosuppressive therapy including systemic or enteric corticosteroids at screening or for the duration of the trial, at the discretion of the site investigator and medical monitor.
7. Use within 5 days prior to randomization or for the duration of the trial of a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4 or expected requirement for chronic use of a strong inhibitor or inducer of CYP3A4 during study therapy.
8. Use within 5 days prior to randomization or for the duration of the trial of drug that is a moderate-to-strong substrate of CYP2C9 (including warfarin, tolbutamide, phenytoin, glimepiride) or expected requirement for chronic use of such drugs during study therapy, at the discretion of the site investigator and medical monitor.
9. Use of investigational treatments for ALS (off-label use or active participation in a clinical trial) within 5 half-lives (if known) or 30 days (whichever is longer) prior to the Screening Visit.
10. Exposure at any time to any gene therapies under investigation for the treatment of ALS (off-label use or investigational).
11. If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or of child-bearing potential and unwilling to use effective contraception for the duration of the trial and for 3 months after discontinuing treatment.
12. If male of reproductive capacity, unwilling to use effective contraception for the duration of the trial and for 3 months after discontinuing study treatment.
13. Anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study, in the SI's opinion.
14. If a participant is being re-screened, the disqualifying condition has not been resolved, or the mandatory wash-out duration has not occurred.
15. Contraindication to undergoing a lumbar puncture (LP) in the SI's opinion. Participants undergoing the LP must not be currently taking anticoagulation and antiplatelet medications such as warfarin and clopidogrel bisulfate (Plavix™), that would be a contraindication to LP; aspirin and non-steroidal anti-inflammatories are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Safety of LAM-002A: occurrence of TEAEs | 28 Weeks
  The occurrence of serious and non-serious treatment-emergent adverse events (TEAEs) and clinically significant treatment-emergent abnormalities in clinical and laboratory values.
Tolerability of LAM-002A: completion of core study treatment | 12 Weeks
  The percentage of participants who complete 12 weeks on study treatment during the Core Study.
Plasma Pharmacokinetics of LAM-002A | 24 Weeks
  The levels of LAM-002 and metabolites in plasma levels.
CSF Pharmacokinetics of LAM-002A | 24 Weeks
  The levels of LAM-002 and metabolites in cerebral spinal fluid (CSF) levels.

SECONDARY OUTCOMES:
Changes in biomarkers | 24 Weeks
  Changes in plasma and CSF levels of a LAM-002A-induced biomarker.
Tolerability of LAM-002A: completion of open-label study treatment | 12 Weeks
  Secondary measures of tolerability will consider completion of 12 weeks on open-label study treatment during the OLE.

OTHER OUTCOMES:
Changes in ALSFRS-R | 28 Weeks
  Change in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) total and domain scores. Score ranges from 0-48 with the higher the score indicating better function.
Changes in Vital Capacity | 24 Weeks
  Change in vital capacity (VC).
Permanent assisted ventilation-free survival | 24 Weeks
  Change in percent of ventilation-free survival summaries.
Changes in ALS-CBS | 24 Weeks
  Change in Amyotrophic Lateral Sclerosis Cognitive Behavioral Scale (ALS-CBS). Comprised of two sub-scores. The cognitive sub-score is rated 0-20 with the higher the score the better patient cognitive function. The caregiver sub-score is rated 0-45 with the higher the score the better patient cognitive function as assessed by their caregiver.
Exploratory biomarkers | 24 Weeks
  Analysis of exploratory disease related biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Suma Babu, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babu S, Nicholson KA, Rothstein JD, Swenson A, Sampognaro PJ, Pant P, Macklin EA, Spruill S, Paganoni S, Gendron TF, Prudencio M, Petrucelli L, Nix D, Landrette S, Nkrumah E, Fandrick K, Edwards J, Young PR. Apilimod dimesylate in C9orf72 amyotrophic lateral sclerosis: a randomized phase 2a clinical trial. Brain. 2024 Sep 3;147(9):2998-3008. doi: 10.1093/brain/awae109. PMID 38606777